CLINICAL TRIAL: NCT02580929
Title: Effectiveness of Radiotherapy Before Surgery in Patients With High-risk Relapse Hepatocellular Carcinoma
Brief Title: Clinical Study of Effectiveness of Radiotherapy Before Surgery in High-risk Relapse Hepatocellular Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Collaborators: Beijing Hope Run (Other)
Responsible Party: Principal Investigator, WU FAN, Doctor, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2014B10
Record Dates: First submitted 2015-10-10; First posted 2015-10-20 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Radiotherapy; General Surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiation (Experimental)
  Interventions: Radiation: radiotherapy
- no radiation (No Intervention)

INTERVENTIONS:
Radiation: radiotherapy — radiotherapy before surgery
  Arms: radiation

SUMMARY:
This study aims to evaluate the effectiveness of radiotherapy before surgery in high-risk relapse hepatocellular cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of HCC
2. In high risk of recurrence of HCC but still can endure palliative resection
3. KPS scores are >90
4. With Child-Pugh Class A liver funcion, serum bilirubin< 1.5*normal maxism; ALT and AST< 1.5*normal maxism; normal creatinine and urea nitrogen; WBC>4×109/L, Hb>110g/L, PLT>90X109/L.
5. Have signed informed consent

Exclusion Criteria:

1. HCC cannot be operated
2. With Child-Pugh Class B/C
3. Have other organ cancer, excluding curative non-melanotic skin cancer and carcinoma in situ of cervix
4. Have other severe disease
5. With active hepatitis
6. Have accepted local radiation therapy in other hospitals
7. KPS scores≤70
8. Tumor edges cannot be defined
9. Have severe cirrhosis complication
10. Intensity modulated radiation therapy cannot reach required dose
11. Cannot cooperate
12. Lactant or pregnant
13. Cannnot be informed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
mortality | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- WU FAN, Beijing, China

REFERENCES:
- [Derived] Wu F, Chen B, Dong D, Rong W, Wang H, Wang L, Wang S, Jin J, Song Y, Liu Y, Fang H, Tang Y, Li N, Zhu X, Li Y, Wang W, Wu J. Phase 2 Evaluation of Neoadjuvant Intensity-Modulated Radiotherapy in Centrally Located Hepatocellular Carcinoma: A Nonrandomized Controlled Trial. JAMA Surg. 2022 Dec 1;157(12):1089-1096. doi: 10.1001/jamasurg.2022.4702. PMID 36197682